CLINICAL TRIAL: NCT01131754
Title: STUDIO CLINICO RANDOMIZZATO SULL'UTILIZZO DI EPARINA PER LA PROFILASSI DELLA TROMBOFLEBITE DA CATETERE VENOSO PERIFERICO
Brief Title: Heparin 100U/L for Prevention of PVC Complications
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Carlo Balduini, Medicina 3 - Fondazione IRCCS Policlinico San Matteo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPA 2007; 2007-001347-21 (EudraCT Number)
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2007-02

CONDITIONS: Peripheral Venous Catheter Complications; Occlusion; Phlebitis; Ecchymosis
Keywords: Peripheral venous catheter complications; PVC occlusion; PVC phlebitis
MeSH Terms: conditions — Bites and Stings; Phlebitis; Ecchymosis | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heparin sol 100U/L (Experimental): peripheral venous catheter flushing with 3 mL of a 100 U heparin/mL normal saline from mono-use vial (Epsodilave, Mayne Pharma, Naples, Italy) at the end of each drug infusion. Independently from the number of drug infusions, all patients will receive at least two catheter flushes every day.
  Interventions: Other: heparin 100U/L flushes
- saline (Active Comparator): peripheral venous catheter flushing with 3 mL of normal saline from mono-use vials (prepared by the hospital pharmacy) at the end of each drug infusion. Independently of the number of drug infusions, all patients will receive at least two catheter flushes every day.
  Interventions: Other: heparin 100U/L flushes

INTERVENTIONS:
Other: heparin 100U/L flushes — peripheral venous catheter flushing with 3 mL of a 100 U heparin/mL normal saline from mono-use vial (Epsodilave, Mayne Pharma, Naples, Italy) at the end of each drug infusion. Independently from the number of drug infusions, all patients will receive at least two catheter flushes every day.

SUMMARY:
Flushes with saline solution are used for maintaining patency of peripheral intermittent intravenous catheters in many institution based on the results of previous studies showing that 10 U heparin/mL is not better than saline in this respect. The latest meta-analysis investigated also safety and efficacy of heparin concentrations of 100 U/ml used as an intermittent flush, but no firm conclusion was reached because of limitations of the few available studies.

ELIGIBILITY:
Inclusion Criteria:

* requiring i.v. therapy for an expected duration longer than five days
* admitted to the 3rd medical ward of IRCCS Policlinico San Matteo

Exclusion Criteria:

* bleeding tendency
* platelet count less than 100 x 109/L
* coagulation defects
* previous adverse reaction to heparin
* programmed cytotoxic therapy
* inability to give an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2007-06; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Phlebitis or Occlusion
  Phlebitis is defined as the presence of two or more symptoms/signs among pain, tenderness, warmth, erythema, swelling, or a palpable cord (score of ≥ 2 according to the Visual Infusion Phlebitis Score). Occlusion is defined as resistance to flushing as evidenced by the inability to administer 1 ml of flushing solution within 30 seconds.

SECONDARY OUTCOMES:
Ecchymosis
  Ecchymosis is defined as a purple discoloration of the skin around the catheter insertion site larger than 1 cm.
Heparin induced thrombocytopenia
  Heparin induced thrombocytopenia is defined as a fall in platelet count > 50% of baseline value without any alternative explanation. To detect this phenomenon, platelet count is to be performed at baseline and, subsequently, every 5 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Medicina 3 - IRCCS Policlinico San Matteo, Pavia, Italy